CLINICAL TRIAL: NCT04597489
Title: Fractional FLOw Reserve In Cardiovascular DiseAses
Acronym: FLORIDA
Status: Completed | Type: Observational
Sponsor: LinkCare GmbH (Industry)
Collaborators: Abbott (Industry); Charite University, Berlin, Germany (Other); University Hospital, Zürich (Other); University Hospital Schleswig-Holstein (Other); Ruhr University of Bochum (Other)
Responsible Party: Sponsor
Other Study IDs: VF/1021/1084
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome | interventions — Fractional Flow Reserve, Myocardial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Angiography + FFR: Patients were stratified into the FFR group if a coronary angiography with adjunctive FFR measurement was performed during the index hospitalization.
  Interventions: Procedure: Fractional flow reserve
- Angiography only: Patients were stratified into the angiography-only group if a coronary angiography without adjunctive FFR measurement was performed.
  Interventions: Procedure: Angiography-only
- Subgroup ACS: Patients were stratified by index diagnoses, i.e. acute coronary syndrome (ACS) or chronic coronary syndrome (CCS) according to the index hospital admission diagnosis.
  This subgroup consists of patients presenting with ACS.
  Interventions: Procedure: Fractional flow reserve; Procedure: Angiography-only
- Subgroup CCS: Patients were stratified by index diagnoses, i.e. acute coronary syndrome (ACS) or chronic coronary syndrome (CCS) according to the index hospital admission diagnosis.
  This subgroup consists of patients presenting with CCS.
  Interventions: Procedure: Fractional flow reserve; Procedure: Angiography-only
- Subgroup revascularization: Patients were stratified by the type of treatment, i.e. percutaneous coronary intervention (PCI), coronary artery bypass grafting (CABG), or conservative management with optimal medical therapy (OMT) alone, based on the procedure codes during the index hospital stay.
  This subgroup consists of patients undergoing revascularization after an angiography (with or without FFR) during the index hospital stay.
  Interventions: Procedure: Fractional flow reserve; Procedure: Angiography-only
- Subgroup optimal medical therapy: Patients were stratified by the type of treatment, i.e. percutaneous coronary intervention (PCI), coronary artery bypass grafting (CABG), or conservative management with optimal medical therapy (OMT) alone, based on the procedure codes during the index hospital stay.
  This subgroup consists of patients undergoing optimal medical therapy after an angiography (with or without FFR) during the index hospital stay.
  Interventions: Procedure: Fractional flow reserve; Procedure: Angiography-only

INTERVENTIONS:
Procedure: Fractional flow reserve — Patients were stratified into the FFR group if a coronary angiography with adjunctive FFR measurement was performed during the index hospitalization.
  Other Names: FFR
  Groups: Angiography + FFR; Subgroup ACS; Subgroup CCS; Subgroup optimal medical therapy; Subgroup revascularization
Procedure: Angiography-only — Patients were stratified into the angiography-only group if a coronary angiography without adjunctive FFR measurement was performed.
  Groups: Angiography only; Subgroup ACS; Subgroup CCS; Subgroup optimal medical therapy; Subgroup revascularization

SUMMARY:
The FLORIDA (Fractional FLOw Reserve In cardiovascular DiseAses) study sought to investigate outcomes of FFR-guided versus angiography-guided treatment strategies in a large, real-world cohort.

DETAILED DESCRIPTION:
The objective of the FLORIDA study was to investigate mortality outcomes of FFR-guided versus angiography-guided treatment strategies in a large, real-world patient cohort, including patients with different stages of coronary artery disease as well as patients with acute coronary syndrome (ACS). All patients were followed for a period of 3 years after the index date. The analysis period extended from the individual index date to the date of death or the end of the 3-year follow-up period. Patients were matched for sex, presence of acute coronary syndrome, age ± 5 years, and propensity scores estimated with logistic regression based on 72 variables , with each FFR patient matched to the closest angiography-only patient

ELIGIBILITY:
Inclusion Criteria:

* At least one inpatient coronary angiography for suspected coronary artery disease between January 2014 and December 2015.

Exclusion Criteria:

* Loss to follow-up of other reasons than death (i.e. change of insurance)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Out of a dataset of 4,395,540 anonymized age- and sex-stratified people from an anonymized German health claims database, patients undergoing at least one inpatient coronary angiography for suspected coronary artery disease between January 2014 and December 2015 were included in the analysis. The discharge date of the first hospital stay involving a coronary angiography was defined as the patient's individual index date. Patients were included into the study population regardless of their underlying disease (all-comers approach), if they were observable for at least four years (one year prior the time of inclusion and three years after the time of inclusion), or died within follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 64045 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 36 months
  All patients were followed for a period of 3 years after the index date. The analysis period extended from the individual index date to the date of death or the end of the 3-year follow-up period. The primary endpoint was mortality at 3 years, prospectively assessed at a quarterly basis.

SECONDARY OUTCOMES:
All-cause mortality | 12 months
  Prospectively assessed at a quarterly basis.
All-cause mortality | 24 months
  Prospectively assessed at a quarterly basis.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Vogelmann, MSc, Study Chair — LinkCare GmbH
Locations (1):
- LinkCare GmbH, Stuttgart, Germany

IPD SHARING:
Plan to Share IPD: No